CLINICAL TRIAL: NCT05064800
Title: A PHASE 1, OPEN-LABEL, 3-TREATMENT, 6-SEQUENCE, 3-PERIOD CROSSOVER STUDY TO ESTIMATE THE EFFECT OF PF-07321332/RITONAVIR AND RITONAVIR ON THE PHARMACOKINETICS OF DABIGATRAN IN HEALTHY PARTICIPANTS
Brief Title: PF-07321332/Ritonavir and Ritonavir on Dabigatran Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671012
Record Dates: First submitted 2021-09-01; First posted 2021-10-01 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-10

CONDITIONS: Healthy Participants
Keywords: Drug Drug Interaction; Dabigatran; P-gp Substrate; SARS-Co-V2; COVID-19; protease inhibitor; ritonavir
MeSH Terms: conditions — COVID-19 | interventions — Dabigatran; nirmatrelvir; Ritonavir

STUDY DESIGN:
Intervention Model Description: This is a Phase1, open-label,3-treatment, 6-sequence, 3-period crossover study to estimate the effect of PF-07321332/ritonavir and ritonavir on the Pharmacokinetics of dabigatran in healthy participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Active Comparator): Dabigatran only
  Interventions: Drug: Dabigatran
- Treatment B (Experimental): PF-07321332/ritonavir + Dabigatran
  Interventions: Drug: PF-07321332/ritonavir + Dabigatran
- Treatment C (Active Comparator): Ritonavir + Dabigatran
  Interventions: Drug: Ritonavir + Dabigatran

INTERVENTIONS:
Drug: Dabigatran — A single dose of Dabigatran on Day 1
  Arms: Treatment A
Drug: PF-07321332/ritonavir + Dabigatran — PF-07321332/ritonavir twice daily (BID) for Days 1 and 2 Single dose of Dabigatran on Day 2
  Arms: Treatment B
Drug: Ritonavir + Dabigatran — Ritonavir BID on Days 1 and 2 Single dose of Dabigatran on Day 2
  Arms: Treatment C

SUMMARY:
This is a drug-drug interaction study to assess the effects of PF-07321332/ritonavir and ritonavir on the Pharmacokinetic (PK) of dabigatran in healthy volunteers. PK will be evaluated for PF-07321332 and ritonavir. Dabigatran is being utilized as a P-gp substrate

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg.m2; and a total body weight >50 kg (110 lbs)
* Female participants must have a negative pregnancy test

Exclusion Criteria:

* Positive test for SARS-Co-V2 at the time of screening or Day -1
* Active pathological bleeding or risk of bleeding
* Positive urine drug test
* History of sensitivity to heparin or heparin induced thrombocytopenia
* Participants who have been vaccinated for COVID-19 in the past 7 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Research Centers of America ( Hollywood ), Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Cox DS, Rehman M, Khan T, Ginman K, Salageanu J, LaBadie RR, Wan K, Damle B. Effects of nirmatrelvir/ritonavir on midazolam and dabigatran pharmacokinetics in healthy participants. Br J Clin Pharmacol. 2023 Nov;89(11):3352-3363. doi: 10.1111/bcp.15835. Epub 2023 Jul 12. PMID 37354048
- [Derived] Sagawa K, Lin J, Jaini R, Di L. Physiologically-Based Pharmacokinetic Modeling of PAXLOVID with First-Order Absorption Kinetics. Pharm Res. 2023 Aug;40(8):1927-1938. doi: 10.1007/s11095-023-03538-5. Epub 2023 May 25. PMID 37231296
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671012

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 24 participants were enrolled into the study, and 4 participants were assigned to each of the 6 sequences to receive following treatments:
  Treatment 1: dabigatran 75 mg orally (PO) single dose Treatment 2: PF-07321332/ritonavir 300 mg/100 mg PO q12h for 2 days + dabigatran 75 mg PO single dose on Day 2 Treatment 3: ritonavir 100 mg PO q12h for 2 days + dabigatran 75 mg PO single dose on Day 2
Groups:
- Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg: For participants in Sequence 1:
  In Period 1, participants received Dabigatran orally as a 75 mg single dose followed by a 3-day washout.(Treatment 1) In Period 2, participants received PF-07321332/ritonavir 300 mg/100 mg every 12 hours (q12h) as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose, followed by a 3-day washout. (Treatment 2) In Period 3, participants received ritonavir 100 mg every 12 hours (q12h) as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose. (Treatment 3)
- Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg: For participants in Sequence 6:
  In Period 1, participants received Dabigatran orally as a 75 mg single dose followed by a 3-day washout.
  In Period 2, participants received ritonavir 100 mg every 12 hours (q12h) as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose.
  In Period 3, participants received PF-07321332/ritonavir 300 mg/100 mg q12h as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose. Treatment 2 was followed by a 3-day washout.
- PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg: For participants in Sequence 5:
  In Period 1, participants received PF-07321332/ritonavir 300 mg/100 mg q12h as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose. Treatment 2 was followed by a 3-day washout.
  In Period 2, participants received Dabigatran orally as a 75 mg single dose followed by a 3-day washout.
  In Period 3, participants received ritonavir 100 mg every 12 hours (q12h) as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose.
- PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg: For participants in Sequence 3:
  In Period 1, Participants received PF-07321332/ritonavir 300 mg/100 mg q12h as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose. Treatment 2 was followed by a 3-day washout.
  In Period 2, Participants received ritonavir 100 mg every 12 hours (q12h) as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose.
  In Period 3, Participants received Dabigatran orally as a 75 mg single dose followed by a 3-day washout.
- Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg: For participants in Sequence 2:
  In Period 1, Participants received ritonavir 100 mg every 12 hours (q12h) as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose.
  In Period 2, Participants received Dabigatran orally as a 75 mg single dose followed by a 3-day washout.
  In Period 3, Participants received PF-07321332/ritonavir 300 mg/100 mg q12h as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose. Treatment 2 was followed by a 3-day washout.
- Ritonavir 100mg+Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg: For participants in Sequence 4:
  In Period 1, Participants received ritonavir 100 mg every 12 hours (q12h) as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose.
  In Period 2, Participants received PF-07321332/ritonavir 300 mg/100 mg q12h as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose. Treatment 2 was followed by a 3-day washout.
  In Period 3, Participants received Dabigatran orally as a 75 mg single dose followed by a 3-day washout.
Period: Period 1
Arm/Group | Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg | Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg | PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg | PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg | Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg | Ritonavir 100mg+Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg | Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg | PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg | PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg | Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg | Ritonavir 100mg+Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg | Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg | PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg | PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg | Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg | Ritonavir 100mg+Dabigatran 75mg=>PF-07321332 300mg+Ritonavir 100mg+Dabigatran 75mg=>Dabigatran 75mg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Groups:
- Enrolled Set: Enrolled set is defined as all participants legally authorized representative's, agreement to participate in this study following completion of the informed consent process and screening.
Arm/Group | Enrolled Set
Number analyzed (Participants) | 24
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0
  18-44 | 9
  45-64 | 15
  >=65 | 0
  Unspecified | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17
  Black or African American | 6
  Asian | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 0
  Unknown | 0
  Multiracial | 1
  Not reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Plasma Dabigatran (Total) PK Parameters (PF-07321332/Ritonavir Co-administered With Dabigatran [Treatment 2]): Maximum Plasma Concentration (Cmax)
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: Treatment 1 Day 1 pre-dose, and at 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose. Treatment 2 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment 1: Dabigatran 75 mg: Dabigatran was administered orally as a 75 mg single dose followed by a 3-day washout.
- Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg: PF-07321332/ritonavir 300 mg/100 mg every 12 hours (q12h) was administered as a multiple dose over a period of 2 days. In the morning on Treatment 2 Day 2, 75 mg of dabigatran was administered orally as a single dose.
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24
ng/mL | 71.87 (78) | 154.1 (72)
Statistical Analysis 1: Comparison: Treatment 1: Dabigatran 75 mg vs Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg; Treatment 1 was Reference and Treatment 2 was Test. Natural log-transformed Cmax of dabigatran was analyzed using mixed effect model with treatment, period, sequence as fixed effects; participant within sequence as a random effect. Estimates of the adjusted mean differences(AMD) (Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Ratio of Adjusted Geometric Means = 233.06, 90% CI 2-sided [172.14 to 315.54]

2. Primary Outcome: Plasma Dabigatran (Total) PK Parameters (PF-07321332/Ritonavir Co-administered With Dabigatran [Treatment 2]): AUCinf
Description: AUCinf was defined as the area under the plasma concentration-time curve from time 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24
ng*hr/mL | 625.6 (61) | 1177 (66)
Statistical Analysis 1: Comparison: Treatment 1: Dabigatran 75 mg vs Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg; Treatment 1 was Reference and Treatment 2 was Test. Natural log-transformed AUCinf of dabigatran was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences(AMD)(Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means(Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Ratio of Adjusted Geometric Means = 169.07, 90% CI 2-sided [135.25 to 211.35]

3. Primary Outcome: Plasma Dabigatran (Total) PK Parameters (PF-07321332/Ritonavir Co-administered With Dabigatran [Treatment 2]): AUClast
Description: AUClast was defined as area under the plasma concentration time curve from time 0 to the time of the last measurable concentration.
Time Frame: as for outcome 1
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24
ng*hr/mL | 595.0 (65) | 1178 (68)
Statistical Analysis 1: Comparison: Treatment 1: Dabigatran 75 mg vs Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg; Treatment 1 was Reference and Treatment 2 was Test. Natural log-transformed AUClast of dabigatran was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences(AMD)(Test-Reference) and 90%CIs were obtained from the model.The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means(Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Ratio of Adjusted Geometric Means = 160.05, 90% CI 2-sided [119.19 to 214.90]

4. Secondary Outcome: Plasma Dabigatran (Total) PK Parameters (Ritonavir Co-administered With Dabigatran [Treatment 3]): Maximum Plasma Concentration (Cmax)
Description: Cmax was defined as maximum observed plasma concentration
Time Frame: Treatment 1 Day 1 pre-dose, and at 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose. Treatment 3 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg: Ritonavir 100 mg q12h was administered as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose.
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24
ng/mL | 71.87 (78) | 117.9 (123)
Statistical Analysis 1: Comparison: Treatment 1: Dabigatran 75 mg vs Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg; Treatment 1 was Reference and Treatment 3 was Test. Natural log-transformed Cmax of dabigatran was analyzed using mixed effect model with treatment, period, sequence as fixed effects; participant within sequence as a random effect. Estimates of the adjusted mean differences(AMD) (Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Ratio of Adjusted Geometric Means = 171.91, 90% CI 2-sided [127.51 to 231.77]

5. Secondary Outcome: Plasma Dabigatran (Total) PK Parameters (Ritonavir Co-administered With Dabigatran [Treatment 3]): AUCinf
Description: AUCinf was defined as area under the plasma concentration-time curve from time 0 extrapolated to infinity
Time Frame: as for outcome 4
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24
ng*hr/mL | 625.6 (61) | 1079 (65)
Statistical Analysis 1: Comparison: Treatment 1: Dabigatran 75 mg vs Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg; Treatment 1 was Reference and Treatment 3 was Test. Natural log-transformed AUCinf of dabigatran was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences(AMD)(Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means(Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Ratio of Adjusted Geometric Means = 169.07, 90% CI 2-sided [135.25 to 211.35]

6. Secondary Outcome: Plasma Dabigatran (Total) PK Parameters (Ritonavir Co-administered With Dabigatran [Treatment 3]): AUClast
Description: as for outcome 3
Time Frame: as for outcome 4
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24
ng*hr/mL | 595.0 (65) | 909.3 (124)
Statistical Analysis 1: Comparison: Treatment 1: Dabigatran 75 mg vs Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg; Treatment 1 was Reference and Treatment 3 was Test. Natural log-transformed AUClast of dabigatran was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences(AMD)(Test-Reference) and 90%CIs were obtained from the model.The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means(Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Ratio of Adjusted Geometric Means = 160.05, 90% CI 2-sided [119.19 to 214.90]

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs , and TEAEs Leading to Participant Discontinuation From Study
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug.
Time Frame: From Pre-dose on Day 1 to Day 48
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg: PF-07321332/ritonavir 300 mg/100 mg q12h was administered as a multiple dose over a period of 2 days. In the morning on Day 2, 75 mg of dabigatran was administered orally as a single dose.
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants
  All-Causality AEs | 3 | 5 | 2
  Treatment-Related AEs | 0 | 2 | 1
  All-Causality SAEs | 0 | 0 | 0
  Treatment-Related SAEs | 0 | 0 | 0
  All-Causality AEs leading to discontinuation from study | 0 | 0 | 0
  Treatment-Related AEs leading to discontinuation from study | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Laboratory Test Abnormality (Without Regard to Baseline Abnormality)
Description: To determine if there are any clinically significant laboratory abnormalities, the haematological, clinical chemistry (serum) and urinalysis safety tests were assessed against the criteria specified in the sponsor reporting standards. Tests including Ery. Mean Corpuscular Hemoglobin, Eosinophils, Activated Partial Thromboplastin Time, Bilirubin, Fibrinogen, URINE Hemoglobin, Nitrite, and Leukocyte Esterase tests.
Time Frame: From pre-dose on Day 1 to Day 3
Population: All participants with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Ery. Mean Corpuscular Hemoglobin (pg/cell) < 0.9x LLN: number analyzed (Participants) | 24 | 23 | 24
  Ery. Mean Corpuscular Hemoglobin (pg/cell) < 0.9x LLN | 1 | 1 | 1
  Eosinophils (10^3/mm^3) > 1.2x ULN: number analyzed (Participants) | 24 | 23 | 24
  Eosinophils (10^3/mm^3) > 1.2x ULN | 1 | 1 | 0
  Activated Partial Thromboplastin Time (sec) > 1.1x ULN: number analyzed (Participants) | 24 | 23 | 24
  Activated Partial Thromboplastin Time (sec) > 1.1x ULN | 0 | 2 | 2
  Bilirubin (mg/dL) > 1.5x ULN: number analyzed (Participants) | 24 | 23 | 24
  Bilirubin (mg/dL) > 1.5x ULN | 1 | 0 | 0
  Fibrinogen (mg/dL) > 1.25x Baseline: number analyzed (Participants) | 24 | 23 | 24
  Fibrinogen (mg/dL) > 1.25x Baseline | 1 | 2 | 1
  URINE Hemoglobin ≥ 1: number analyzed (Participants) | 24 | 23 | 24
  URINE Hemoglobin ≥ 1 | 6 | 6 | 6
  Nitrite ≥ 1: number analyzed (Participants) | 24 | 23 | 24
  Nitrite ≥ 1 | 3 | 3 | 1
  Leukocyte Esterase ≥ 1: number analyzed (Participants) | 24 | 23 | 24
  Leukocyte Esterase ≥ 1 | 4 | 4 | 2

9. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Concern
Description: Single supine blood pressure and pulse rate tests were assessed against the criteria specified in the sponsor reporting standards.
Time Frame: From pre-dose on Day 1 to Day 3
Population: All participants evaluated against criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Systolic Blood Pressure Value < 90 mmHg: number analyzed (Participants) | 24 | 23 | 24
  Systolic Blood Pressure Value < 90 mmHg | 2 | 2 | 0
  Systolic Blood Pressure Change ≥ 30 mmHg increase: number analyzed (Participants) | 24 | 23 | 24
  Systolic Blood Pressure Change ≥ 30 mmHg increase | 0 | 2 | 0
  Systolic Blood Pressure Change ≥ 30 mmHg decrease: number analyzed (Participants) | 24 | 23 | 24
  Systolic Blood Pressure Change ≥ 30 mmHg decrease | 0 | 1 | 0
  Diastolic Blood Pressure Value < 50 mmHg: number analyzed (Participants) | 24 | 23 | 24
  Diastolic Blood Pressure Value < 50 mmHg | 1 | 1 | 0
  Diastolic Blood Pressure Change ≥ 20 mmHg increase: number analyzed (Participants) | 24 | 23 | 24
  Diastolic Blood Pressure Change ≥ 20 mmHg increase | 0 | 1 | 1
  Diastolic Blood Pressure Change ≥ 20 mmHg decrease: number analyzed (Participants) | 24 | 23 | 24
  Diastolic Blood Pressure Change ≥ 20 mmHg decrease | 1 | 2 | 0
  Pulse Rate Value < 40 bpm: number analyzed (Participants) | 24 | 23 | 24
  Pulse Rate Value < 40 bpm | 0 | 0 | 0
  Pulse Rate Value > 120 bpm: number analyzed (Participants) | 24 | 23 | 24
  Pulse Rate Value > 120 bpm | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With ECG Values of Potential Clinical Concern
Description: QT interval, QTc, PR, RR, QRS and heart rate tests were assessed against the criteria specified in the sponsor reporting standards.
Time Frame: From pre-dose on Day 1 to Day 3
Population: All participants evaluated against criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24 | 24 | 24
Participants
  PR Interval not Otherwise Specified Value ≥ 300 MSEC: number analyzed (Participants) | 24 | 23 | 24
  PR Interval not Otherwise Specified Value ≥ 300 MSEC | 0 | 0 | 0
  PR Interval not Otherwise Specified %Change ≥ 25/50%: number analyzed (Participants) | 24 | 23 | 24
  PR Interval not Otherwise Specified %Change ≥ 25/50% | 1 | 0 | 0
  QRS Interval not Otherwise Specified Value ≥ 140 MSEC: number analyzed (Participants) | 24 | 23 | 24
  QRS Interval not Otherwise Specified Value ≥ 140 MSEC | 0 | 0 | 0
  QRS Interval not Otherwise Specified %Change ≥ 50%: number analyzed (Participants) | 24 | 23 | 24
  QRS Interval not Otherwise Specified %Change ≥ 50% | 0 | 0 | 0
  QTCF not Otherwise Specified 450 MSEC ≤ Value < 480 MSEC: number analyzed (Participants) | 24 | 23 | 24
  QTCF not Otherwise Specified 450 MSEC ≤ Value < 480 MSEC | 0 | 0 | 0
  QTCF not Otherwise Specified 480 MSEC ≤ Value < 500 MSEC: number analyzed (Participants) | 24 | 23 | 24
  QTCF not Otherwise Specified 480 MSEC ≤ Value < 500 MSEC | 0 | 0 | 0
  QTCF not Otherwise Specified Value ≥ 500 MSEC: number analyzed (Participants) | 24 | 23 | 24
  QTCF not Otherwise Specified Value ≥ 500 MSEC | 0 | 0 | 0
  QTCF not Otherwise Specified 30 MSEC ≤ Change < 60 MSEC: number analyzed (Participants) | 24 | 23 | 24
  QTCF not Otherwise Specified 30 MSEC ≤ Change < 60 MSEC | 0 | 0 | 0
  QTCF not Otherwise Specified Change ≥ 60 MSEC: number analyzed (Participants) | 24 | 23 | 24
  QTCF not Otherwise Specified Change ≥ 60 MSEC | 0 | 0 | 0

11. Secondary Outcome: Plasma Dabigatran (Total) PK Parameters (PF-07321332/Ritonavir Co-administered With Dabigatran [Treatment 2]): Time to First Occurrence of Cmax (Tmax)
Description: Tmax was defined as time to first occurrence of Cmax
Time Frame: Treatment 2 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
hours | 2.000 [2.00 to 4.00]

12. Secondary Outcome: Plasma Dabigatran (Total) PK Parameters (Ritonavir Co-administered With Dabigatran [Treatment 3]): Tmax
Description: Tmax was defined as time to first occurrence of Cmax.
Time Frame: Treatment 3 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
hours | 2.000 [1.00 to 4.00]

13. Secondary Outcome: Plasma Dabigatran (Total) PK Parameters (PF-07321332/Ritonavir Co-administered With Dabigatran [Treatment 2]): Terminal Half-life (t½)
Description: t½ was defined as terminal half-life of Dabigatran (Total) PK Parameters (PF-07321332/ritonavir co-administered with dabigatran.
Time Frame: Treatment 2 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
hours | 9.636 (1.5692)

14. Secondary Outcome: Plasma Dabigatran (Total) PK Parameters (Ritonavir Co-administered With Dabigatran [Treatment 3]): t½
Description: t½ was defined as terminal half-life of Dabigatran (Total).
Time Frame: Treatment 3 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
hours | 10.16 (1.3350)

15. Secondary Outcome: Plasma PF-07321332 PK Parameters: Cmax
Time Frame: Treatment 2 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
ng/mL | 4065 (76)

16. Secondary Outcome: Plasma PF-07321332 PK Parameters: AUCtau
Description: AUCtau was defined as area under the plasma concentration-time profile from time zero to time tau (τ) the dosing interval, where tau=12 hours for twice daily (BID) dosing.
Time Frame: Treatment 2 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
ng*hr/mL | 30080 (78)

17. Secondary Outcome: Plasma PF-07321332 PK Parameters: t½
Description: t½ was defined as terminal half-life of PF-07321332.
Time Frame: Treatment 2 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
hours | 3.969 (0.53736)

18. Secondary Outcome: Plasma PF-07321332 PK Parameters: Tmax
Description: Tmax was defined as time to first occurrence of Cmax.
Time Frame: Treatment 2 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Mean (Full Range); unit: hours
Arm/Group | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
hours | 2.000 [1.00 to 4.00]

19. Secondary Outcome: Plasma PF-07321332 PK Parameters: CL/F
Description: CL/F was defined as apparent clearance of drug from plasma.
Time Frame: Treatment 2 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
L/hr | 9.975 (78)

20. Secondary Outcome: Plasma PF-07321332 PK Parameters: Vz/F
Description: Vz/F was defined as apparent volume of distribution.
Time Frame: Treatment 2 Day 2 pre-dose, and at 1, 2, 4, 6, 8, 12 hours post-dose
Population: All participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg
Number analyzed (Participants) | 24
Liters | 56.48 (29)

ADVERSE EVENTS:
Time Frame: From Study Day 1 up to Study Day 48
Description: Same event may appear as adverse event (AE) and serious AE, what is presented as distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who were randomized and received at least 1 confirmed dose of investigational product.
Arm/Group | Treatment 1: Dabigatran 75 mg | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 1/24 | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1: Dabigatran 75 mg (N=24) | Treatment 2: PF-07321332 300 mg + Ritonavir 100 mg + Dabigatran 75 mg (N=24) | Treatment 3: Ritonavir 100 mg + Dabigatran 75 mg (N=24)
Headache (Nervous system disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT05064800/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT05064800/SAP_001.pdf